CLINICAL TRIAL: NCT01838733
Title: Cerebral Oximetry and Perioperative Outcome in Non-Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Anesthesia Research Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. Duane Funk, Assistant Professor, University of Manitoba
Other Study IDs: B2013:015
Record Dates: First submitted 2013-04-20; First posted 2013-04-24 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: High Risk Non-cardiac Surgery; Death; Delirium; Kidney Injury; Myocardial Infarction; Respiratory Failure; Postoperative Infection
MeSH Terms: conditions — Death; Delirium; Myocardial Infarction; Respiratory Insufficiency | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebral Desaturation: Patients who suffer an intra-operative cerebral desaturation
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study

SUMMARY:
Cerebral desaturations occur frequently in patients undergoing non-cardiac surgery. The definition of what constitutes a cerebral desaturation, the incidence of the phenomenon, the association between desaturations and perioperative outcome, and the mechanistic explanations of cerebral desaturations remain unexamined. This study seeks to identify the true incidence and magnitude of cerebral desaturations in high-risk non-cardiac surgical patients and the association between desaturations and perioperative outcome.

The investigators will attempt to determine the following (1) The proper definition, incidence and severity of decreased cerebral saturation (rSO2) in high-risk non-cardiac surgical patients (2) the mechanisms surrounding decreases in rSO2 by correlating it with alterations in physiologic parameters (such as blood pressure, cardiac output, hemoglobin concentration, and carbon dioxide levels) and (3) to correlate the incidence and severity of decreased rSO2 with relevant perioperative.

The investigators will also analyze a panel of inflammatory biomarkers to determine if these biomarkers have the ability to predict postoperative complications.

The investigators will study 200 high-risk patients undergoing high-risk non-cardiac surgery. The investigators will determine the incidence and severity of decreases in rSO2, the associated factors with the occurrence of decreased rSO2, and the relationship between decreases in rSO2 and adverse perioperative outcome with a composite of well defined perioperative complications such as death, myocardial infarction, cerebrovascular accident, acute kidney injury, delirium, postoperative infections, and the need for mechanical ventilation.

DETAILED DESCRIPTION:
There have been a number of studies that have examined a link between intraoperative decreases in rSO2 and adverse perioperative outcome3-7. These studies, the vast majority of which have been in the setting of cardiac surgery, suggest that decreases in rSO2 (as detected by near-infrared spectroscopy) may be related to both adverse neurologic and non-neurologic sequelae. Interestingly, and importantly, the studies examining cerebral desaturation in non-cardiac surgical patients (such as those undergoing major abdominal surgery, carotid endarterectomy, liver transplantation, and pulmonary resection) have also uncovered a link between cerebral desaturation and non-neurologic outcomes3,7-12. These small studies have reported preliminary correlates between decreases in rSO2 and various postoperative complications and prolonged length of stay. These studies have also shown that the changes in rSO2 are not correlated with changes in traditional hemodynamic parameters (mean arterial pressure (MAP) and heart rate).

All of these studies suffer from similar flaws, however. They are typically small in size, have varying definitions of what constitutes a cerebral desaturation event, and have incompletely, or poorly defined complications. Also lacking is a mechanistic explanation for the cerebral desaturations as peripheral oxygen saturation typically remains near normal.

As a result, two natural questions arise in relation to this prior research. First, are these cerebral desaturations causative of the adverse outcomes (including non-neurologic complications), and second if these desaturations were treated (i.e. if cerebral oxygenation was normalized) would outcome be improved (i.e. or are cerebral desaturations merely an epiphenomenon)? Numerous studies have demonstrated the poor correlation of traditional hemodynamic parameters (such as blood pressure and heart rate) to cardiac output and oxygen delivery13-17. Historically in the fields of anesthesiology and critical care, we have focused our monitoring and resuscitation targets on perfusion pressures rather than organ flows. Neglecting the fact that organs require flow as well as pressure has led to an over-reliance on normal vascular pressures (such as arterial, central venous, and pulmonary capillary wedge pressures) as a surrogate for adequate organ flow18.

It is entirely possible that monitoring cerebral oxygenation and discovering a link between desaturation and non-neurologic outcomes may show that the brain is an index organ for tissue perfusion monitoring. That is to say, since the perfusion of major organs are typically not monitored during anesthesia, cerebral oximetry is an excellent means to monitor global decreases in tissue oxygen delivery. Consistent with this hypothesis, in the largest cerebral oximetry trial to date, Murkin and colleagues discovered that the incidence and magnitude of cerebral desaturations was related to major non-neurologic organ morbidity19.

The investigators will also be collecting blood samples preoperatively and at 24 hours postoperatively to determine if a panel of inflammatory biomarkers has the ability to predict postoperative complications.

Primary Objective: to determine the incidence and severity of cerebral desaturation in high-risk patients undergoing major vascular and abdominal surgery

Secondary Objectives:

1. To determine the factors associated with the occurrence of cerebral desaturation
2. To determine the relationship between desaturation and adverse perioperative outcome
3. To determine if the levels of a panel of inflammatory biomarkers is related to cerebral desaturation and postoperative complications.

Study design: prospective observational study Population: 200 consecutive high-risk patients undergoing non-cardiac surgery. High-risk patients will be defined as age> 65 undergoing major non-cardiac surgery including abdominal aortic aneurysm repair, major hepatic resection, colonic resection, pancreatoduodenectomy, or esophagectomy.

Methods: In addition to standard CAS monitors, all patients will undergo pulse contour cardiac output monitoring and cerebral oxygen saturation monitoring. The anesthetic technique will be at the discretion of the attending anesthesiologist. During the procedure, the attending anesthesiologist will be blinded to the rSO2 data.

As with previous studies conducted at our institution, cardiorespiratory variables (such as heart rate, systolic, diastolic and mean arterial blood pressures, peripheral and cerebral oxygen saturation, end tidal CO2 tension, end tidal anesthetic gas concentration, and cardiac index) will be sampled at a frequency of 60Hz. Data will be acquired from the Philips Intellivue® Monitor (Philips Healthcare, Andover, MA), FloTrac/Vigileo® minimally invasive CO monitor (Edwards Lifesciences, Orange County, CA), and the ForeSight® Cerebral Oximiter (CasMED, Brantford CT) and processed with TrendFace Solo® software (IExcellence Software, Germany). Arterial blood gas sampling will occur every 20 minutes. Other intraoperative variables collected will include case duration, blood loss, total narcotic dose, total benzodiazepine dose, use and dose of vasopressors, and use of neuraxial local anesthetics.

The definition of a cerebral desaturation differs between previously performed studies. Some have used an absolute decrease below 55%, variably defined decreases from the patients 'baseline' (either breathing room air or 100% oxygen), the time below a specific cerebral saturation threshold, or area under a specific cerebral saturation threshold (this measurement takes into account the duration and magnitude of a desaturation)3,5,21,22. Based on the intraoperative data collected, The investigators will examine all of the currently utilized definitions of cerebral desaturation and then construct receiver operating characteristic curves to determine which parameter has then highest predictive ability to link cerebral desaturation with perioperative outcome.

In consultation with our Biostatistical Consulting Unit the investigators calculated our sample size using previously reported incidences of cerebral desaturation, which range from 15-26% and accepted a margin of error of 5%. Based on a conservative estimate of the incidence (15%), The investigators would need a total of 195 patients to determine the incidence of cerebral desaturations with a 5% margin of error (see figure 1). The investigators will include 5 additional patients in our study due to our previous experience of a 1% rate of data loss during acquisition of rSO2 data (related to technical failures). The Lan and DeMets alpha spending function will be utilized to determine if the trial can be stopped early.

As secondary outcomes, the investigators will attempt to correlate decreases in rSO2 with a composite of well defined perioperative complications such as death, myocardial infarction, cerebrovascular accident, acute kidney injury (defined by the AKIN criteria, table 223), delirium (as defined by the CAM-ICU method, figure 324), postoperative infections, and the need for mechanical ventilation >24 hours in the first 28 postoperative days.

Based on the results of this study the investigators will be able to determine, with the aid of multivariate logistical regression analysis and the calculation of odds ratios, which definition of cerebral desaturation is mostly closely linked with the aforementioned outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age >65
* High risk surgery (aortic aneurysm repair, hepatic resection, pancreatectomy, colon resection)

Exclusion Criteria:

* Previous stroke
* Dementia

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Age >65 High-risk non-cardiac surgery (aortic aneurysm repair, hepatic resection, pancreatectomy, colon resection)
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2014-04; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Cerebral desaturation | Intraoperative

SECONDARY OUTCOMES:
Composite outcome of adverse peri-operative outcome | 28 days
  Death, myocardial infarction, cerebrovascular accident, acute kidney injury (defined by the AKIN criteria), delirium (as defined by the CAM-ICU method), postoperative infections, and the need for mechanical ventilation >24 hours in the first 28 postoperative days.
Levels of perioperative inflammatory biomarkers | 24 Hours
  Levels of a panel of inflammatory biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Duane J Funk, MD FRCP(C), Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Center, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Apostolidou I, Morrissette G, Sarwar MF, Konia MR, Kshettry VR, Wahr JA, Lobbestael AA, Nussmeier NA. Cerebral oximetry during cardiac surgery: the association between cerebral oxygen saturation and perioperative patient variables. J Cardiothorac Vasc Anesth. 2012 Dec;26(6):1015-21. doi: 10.1053/j.jvca.2012.07.011. Epub 2012 Sep 18. PMID 22995459
- [Background] Bellomo R, Ronco C, Kellum JA, Mehta RL, Palevsky P; Acute Dialysis Quality Initiative workgroup. Acute renal failure - definition, outcome measures, animal models, fluid therapy and information technology needs: the Second International Consensus Conference of the Acute Dialysis Quality Initiative (ADQI) Group. Crit Care. 2004 Aug;8(4):R204-12. doi: 10.1186/cc2872. Epub 2004 May 24. PMID 15312219
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Danelli G, Fierro G, De Cosmo G, Servillo G; Collaborative Italian Study Group on Anesthesia in Elderly Patients. Continuous monitoring of cerebral oxygen saturation in elderly patients undergoing major abdominal surgery minimizes brain exposure to potential hypoxia. Anesth Analg. 2005 Sep;101(3):740-747. doi: 10.1213/01.ane.0000166974.96219.cd. PMID 16115985
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Montanini S; Collaborative Italian Study Group on Anaesthesia in Elderly Patients; Danelli G, Nuzzi M, Mentegazzi F, Torri G, Martani C, Spreafico E, Fierro G, Pugliese F, De Cosmo G, Aceto P, Servillo G, Monaco F. Monitoring cerebral oxygen saturation in elderly patients undergoing general abdominal surgery: a prospective cohort study. Eur J Anaesthesiol. 2007 Jan;24(1):59-65. doi: 10.1017/S0265021506001025. Epub 2006 Jul 7. PMID 16824246
- [Background] Casati A, Spreafico E, Putzu M, Fanelli G. New technology for noninvasive brain monitoring: continuous cerebral oximetry. Minerva Anestesiol. 2006 Jul-Aug;72(7-8):605-25. English, Italian. PMID 16865080
- [Background] Colak Z, Borojevic M, Ivancan V, Gabelica R, Biocina B, Majeric-Kogler V. The relationship between prolonged cerebral oxygen desaturation and postoperative outcome in patients undergoing coronary artery bypass grafting. Coll Antropol. 2012 Jun;36(2):381-8. PMID 22856219
- [Background] Davie SN, Grocott HP. Impact of extracranial contamination on regional cerebral oxygen saturation: a comparison of three cerebral oximetry technologies. Anesthesiology. 2012 Apr;116(4):834-40. doi: 10.1097/ALN.0b013e31824c00d7. PMID 22343469
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Green DW. A retrospective study of changes in cerebral oxygenation using a cerebral oximeter in older patients undergoing prolonged major abdominal surgery. Eur J Anaesthesiol. 2007 Mar;24(3):230-4. doi: 10.1017/S0265021506001645. Epub 2006 Oct 23. PMID 17054814
- [Background] Hoppenstein D, Zohar E, Ramaty E, Shabat S, Fredman B. The effects of general vs spinal anesthesia on frontal cerebral oxygen saturation in geriatric patients undergoing emergency surgical fixation of the neck of femur. J Clin Anesth. 2005 Sep;17(6):431-8. doi: 10.1016/j.jclinane.2004.09.013. PMID 16171663
- [Background] Kwak HJ, Park SK, Lee KC, Lee DC, Kim JY. High positive end-expiratory pressure preserves cerebral oxygen saturation during laparoscopic cholecystectomy under propofol anesthesia. Surg Endosc. 2013 Feb;27(2):415-20. doi: 10.1007/s00464-012-2447-5. Epub 2012 Jun 30. PMID 22752286
- [Background] Lee A, Kim SH, Hong JY, Hwang JH. Effect of anesthetic methods on cerebral oxygen saturation in elderly surgical patients: prospective, randomized, observational study. World J Surg. 2012 Oct;36(10):2328-34. doi: 10.1007/s00268-012-1676-z. PMID 22736340
- [Background] Meng L, Cannesson M, Alexander BS, Yu Z, Kain ZN, Cerussi AE, Tromberg BJ, Mantulin WW. Effect of phenylephrine and ephedrine bolus treatment on cerebral oxygenation in anaesthetized patients. Br J Anaesth. 2011 Aug;107(2):209-17. doi: 10.1093/bja/aer150. Epub 2011 Jun 3. PMID 21642644
- [Background] Morimoto Y, Yoshimura M, Utada K, Setoyama K, Matsumoto M, Sakabe T. Prediction of postoperative delirium after abdominal surgery in the elderly. J Anesth. 2009;23(1):51-6. doi: 10.1007/s00540-008-0688-1. Epub 2009 Feb 22. PMID 19234823
- [Background] Paarmann H, Heringlake M, Heinze H, Hanke T, Sier H, Karsten J, Schon J. Non-invasive cerebral oxygenation reflects mixed venous oxygen saturation during the varying haemodynamic conditions in patients undergoing transapical transcatheter aortic valve implantation. Interact Cardiovasc Thorac Surg. 2012 Mar;14(3):268-72. doi: 10.1093/icvts/ivr102. Epub 2011 Dec 7. PMID 22159266
- [Derived] Pries PJ, Mutch WAC, Funk DJ. Characterizing drivers of change in intraoperative cerebral saturation using supervised machine learning. J Clin Monit Comput. 2025 Jun;39(3):559-569. doi: 10.1007/s10877-025-01265-3. Epub 2025 Feb 7. PMID 39920503